CLINICAL TRIAL: NCT03659539
Title: Evaluation of Quality of Recovery With QoR-15 Score Following Closed-Loop Anaesthesia Delivery System Guided Propofol Versus Desflurane General Anaesthesia in Patients Undergoing Transabdominal Robotic Surgery: A Randomized Controlled Study
Brief Title: Quality of Recovery After Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitin Sethi, DNB (Other)
Responsible Party: Sponsor-Investigator, Nitin Sethi, DNB, Associate Professor & Consultant, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/08/18/1393
Record Dates: First submitted 2018-09-02; First posted 2018-09-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Patients Undergoing Robotic Surgery
Keywords: propofol; desflurane; robotic; recovery
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Intervention Model Description: 120-patients aged 18-65 years, ASA physical status I/II, of either sex, and undergoing elective major robotic surgery will be randomly allocated to one of the following two groups:
  Group-1 [CLADS Group, n=60]: Anaesthesia will be induced and maintained with propofol administered using the BIS feedback-based automated CLADS.
  Group-2 [Desflurane Group, n=60]: Anaesthesia will be induced with propofol CLADS and will be maintained intraoperatively by Desflurane titrated to BIS monitoring.
Who Masked: Participant, Outcomes Assessor
Masking Description: The attending anaesthesiologist will not be blinded to the technique utilized to administer GA and also to the in-OR recovery profile immediately after tracheal extubation. However, they will be blinded to postoperative recovery parameters, which will be noted by an independent assessor unaware of the technique utilized for administering GA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLADS group (Active Comparator): Anesthesia will be induced with propofol administered using automated closed loop anesthesia delivery system (CLADS) which will be set to deliver Propofol. A BIS-value of 50 will be used as the target for induction of anesthesia. Thereafter anesthesia maintenance will be done with propofol, with its administration controlled with CLADS tuned to consistent anesthetic depth (BIS-50) feedback from the patients.
  Interventions: Drug: PROPOFOL
- Desflurane group (Active Comparator): Anesthesia will be induced with propofol administered using automated closed loop anesthesia delivery system (CLADS) which will be set to deliver Propofol. A BIS-value of 50 will be used as the target for induction of anesthesia. Thereafter anesthesia maintenance will be done with desflurane using an agent specific vaporiser, whose dial concentration will be adjusted to maintain a BIS of 50-55 in all the patients
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: PROPOFOL — Propofol delivery will be controlled using automated closed loop anaesthesia delivery system which will control propofol delivery rate to consistent anaesthetic depth (BIS-50) feedback from the patient.
  Arms: CLADS group
Drug: Desflurane — Desflurane delivery will be controlled using a agent specific vaporiser. The dial concentration of the vaporiser will be adjusted to maintain a BIS of 50-55 in the patients.
  Arms: Desflurane group

SUMMARY:
Robotic approach to laparoscopic surgery has greatly facilitated undertaking complex surgery inside the abdominal cavity with ease. Robotic surgery is performed under general anaesthesia (GA), which is commonly administered either via the inhalational route or intravenous route. Currently, there is paucity of evidence regarding comprehensive patient outcome following robotic transabdominal surgery. The limited data that is available is restricted to specific outcome parameters such as hemodynamic profile, recovery times, and concomitant effects (post-operative nausea vomiting, pain). QoR (quality of recovery)-15 is a patient self- reported measurement of outcome to assess postoperative QoR. QoR-15 is a15-item questionnaire that assess physical and mental well-being of the patient after anesthesia and surgery. It is the first validated outcome assessment scale that has been evaluated using the Consensus-based Standards for the Selection of health Measurements Instruments (COSMIN) and fulfils the requirements for assessing QoR postoperatively. We plan to conduct this randomized controlled-trial to evaluate postoperative QoR using the QoR-15 questionnaire in patients undergoing robotic abdominal surgery under GA administered by routine techniques, namely, closed-loop anesthesia delivery system (CLADS) controlled total intravenous anesthesia (TIVA) with propofol or inhalation anesthesia with desflurane.

DETAILED DESCRIPTION:
The advent of robotic approach to laparoscopic surgery has transformed the practice of transabdominal procedures, especially those involving the pelvic region, such as, prostatectomy, hysterectomy, among others. In-line with the advantages of robotic intervention (greater access and precision), the type of patients who can undergo this surgery has also evolved. Whereas, morbidly obese patients, who were not amenable to 'open' or even 'laparoscopic' approach because of technical difficulties of gaining access to the operative organ/area; can now safely undergo surgery because of high-fidelity and intuitive robotic instrumentation. However, the robotic technique has its own share of concerns: first, it is difficult for the anesthesiologists to access the patient once the robotic arms are docked in position; and second, the extreme positioning (steep Trendelenberg, anti-Trendelenberg position) required to successfully apply the technique may lead to undue burden/adversity on patient's cardiovascular (tachycardia, hypertension, hypotension), respiratory (decreased lung compliance), and central nervous (elevated intracranial pressures) systems.

Therefore, general anesthesia (GA) techniques employed for robotic surgery should be robust and consistent. The common GA techniques, i.e. inhalational or a total intravenous anesthesia (TIVA) can be used. Advantage of inhalation anesthesia is easy titration of the agent by finely calibrated dial concentration control. In addition, the commonly used inhalation anesthetics such as sevoflurane or desflurane rapidly achieve anesthetic brain concentration and the effect can be efficiently reversed quickly upon discontinuation at the end of surgery. TIVA with intravenous anesthetic like propofol is delivered by via simple or target-controlled infusion pumps. Emerging evidence supports the use of propofol TIVA for it may also proffer decreased incidence of postoperative nausea-and-vomiting, anti-inflammatory effect, and anti-neoplastic action.

The evidence on beneficial effect of prolonged robotic surgery on postoperative patient recovery are scanty, unstructured, and limited only to male patients undergoing radical prostatectomy. For the want of a comprehensive patient assessment protocol, the available outcome study has been able to focus on a limited number of parameters, including, changes in intraocular pressure and the incidence of PONV/postoperative pain. Therefore, for knowing the actual outcome effect of GA for robotic surgery, it is essential to analyze elaborate quality-of-recovery from anesthesia based on compendious patients experiences rather than concentrating on specific end-points (hemodynamic profile, recovery time, etc.).

Quality of recovery-15 (QoR-15), a comprehensive patient-reported measure of quality of post-anesthesia, is an abridged form of the expansive 40-item questionnaire (QoR-40) score. QoR-15 assesses both physical and mental well-being of the patient after surgery under GA and is easier to administer. QoR-15 is the first outcome assessment scale which has been evaluated and validated using the consensus-based standards for the selection of health measurements instruments (COSMIN) and fulfils the requirement for being an effective tool for assessment of postoperative recovery/outcome in clinical trials.

Since there is a paucity of evidence on comprehensive post-anesthesia outcome following major robotic procedures and the choice of GA techniques employed for such procedures are subject to random selection; we aim to undertake this randomized-controlled trial to assess postoperative QoR with QoR-15 questionnaire in patients receiving anesthesia either by propofol administration facilitated by automated closed-loop anesthesia delivery system (CLADS) or desflurane inhalation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I/II
* Undergoing elective robotic surgery of more than 60-minutes duration

Exclusion Criteria:

* Uncompensated cardiovascular illness (uncontrolled hypertension, atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced left ventricular compliance and diastolic dysfunction)
* Pre-existent neurological issues (previous neurosurgical intervention, psychiatric disease, morbid autonomic nervous system: orthostatic hypotension, transient ischemic attacks, history of alcohol/substance abuse, among others)
* Hepato-renal insufficiency
* Endocrinology problems, e.g. uncontrolled diabetes mellitus, hypothyroidism
* Known allergy/hypersensitivity to the study drugs (propofol, desflurane)
* Pulmonary dysfunction (chronic restrictive /obstructive lung disease, chronic smokers)
* Nutritional ailments: obesity (BMI > 30 kg/m2), malnutrition (severe anaemia [Hb < 8gm%] , hypoalbuminemia [< 3.5gm%], bed-ridden moribund status)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Quality-of-recovery | From one day before surgery till postoperative day two
  Quality-of-recovery will be assessed using QoR-15 questionnaire

SECONDARY OUTCOMES:
Anaesthesia depth consistency | From beginning of anesthesia (0-hours, baseline) till 8 hours intraoperatively
  Comparison of anaesthesia depth adequacy using Varvel criteria parameters: percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS (50), median performance error (MDPE), median absolute performance error (MDAPE), and global score
Changes in intra-operative heart rate (beats per minute) | From beginning of anesthesia (0-hours, baseline) till 8 hours intraoperatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative blood pressure - systolic , diastolic, and mean (mmHg) | From beginning of anesthesia (0-hours, baseline) till 8 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Early recovery | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative Sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale (OASS). It is a 6 point scale from 0 (fully sedated) to 5 (fully awake)
Postoperative Nausea and Vomiting | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using PONV Scale. It is a 3 point scale from 0 (no nausea & vomiting) to 2 (vomiting present)
Postoperative Analgeisa | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using 10-point numeric rating scale (NRS). It is a 10 point scale from 0 (no pain) to 10 (maximum pain).
Intra-operative awareness | From the end of anaesthesia till 48-hours postoperatively
  Will be assessed using modified brice questionnaire. It consists of 5 questions pertaining to assessment of intraoperative awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Jayashree Sood, MD, FFRCA, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Goverdhan D Puri, MD, PhD, Study Director — Post Graduate Institute of Medical Education & Research, Chandigarh, India
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No